CLINICAL TRIAL: NCT05748912
Title: Lung Function Outcomes Following Removal of Airway Mucus Plugs in Patients With Asthma
Brief Title: Lung Function Outcomes Following Removal of Airway Mucus Plugs in Patients With Asthma (FOCUS)
Acronym: FOCUS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants were enrolled in protocol A due to COVID-related restrictions and funding issues.
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-33420; 2P01HL107202-06A1 (NIH)
Record Dates: First submitted 2022-01-29; First posted 2023-03-01 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: FOCUS protocol A is a single-arm study which means all study participants will receive the same intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapeutic bronchoscopy for removal of mucus plugs (Experimental): Protocol A: This protocol will study 10 patients with asthma who have CT (Computed Tomography) evidence of mucus plugs in their airways. Screening data will be reviewed to determine participant eligibility. Participants who meet all eligibility criteria will participate in a bronchoscopy done on one lung for the first 5 participants, and if single lung mucus removal is well tolerated then we will perform bronchoscopies on both lungs for the next 5 participants.
  Interventions: Procedure: Therapeutic bronchoscopy for removal of mucus plugs

INTERVENTIONS:
Procedure: Therapeutic bronchoscopy for removal of mucus plugs — Research participants that meet the study inclusion criteria will undergo a research bronchoscopy to remove airway mucus plugs from 1 lung for the first 5 participants, and, if single lung mucus removal is well tolerated, on both lungs for the next 5 participants.

SUMMARY:
This is a single-center study that will evaluate the safety and tolerability of removal of mucus plugs by bronchoscopy in patients with asthma. This protocol will also plan for the analysis of the features of the mucus plugs removed.

DETAILED DESCRIPTION:
The investigators' research shows that a large subgroup of asthma patients have mucus plugs, and quantification of these plugs using a bronchopulmonary segment-based scoring system reveals a strong negative correlation between the CT (Computed Tomography) mucus plug score and FEV1 (Forced Expiratory Volume at 1 second). The FOCUS study is a single-center study that has the overarching goal to explore the biology of airway mucus plugs in asthma.

Through the FOCUS study, the investigators will initially explore the safety and tolerability of bronchoscopic removal of airway mucus plugs in patients with asthma and mucus plugs. They will then evaluate potential improvements in lung function outcomes in a dose-dependent manner (i.e., by removing mucus plugs from one lung vs both lungs). A secondary objective of the FOCUS study is to perform detailed cellular and molecular analyses of mucus and epithelial cells from airways impacted with mucus. With these biospecimens, the investigators intend to extend their preliminary findings that mucus plugged airways are characterized by intense type 2 inflammation, determine the mechanisms of epithelial and immune cell reprogramming, as well as how cellular reprogramming affects the promotion and persistence of type 2 airway inflammation.

ELIGIBILITY:
Protocol A:

Inclusion Criteria:

* Males or females between the ages 18 to 70 at the time of visit 1.
* Clinical history of asthma per patient report or medical record.
* Pre-bronchodilator FEV1 < 80% predicted and ≥ 35% predicted
* CT mucus plug score > 5.
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Smoking of tobacco or other recreational inhalants in the last month and/or >10 pack-year smoking history.
* History of other pulmonary disorders including cystic fibrosis and COPD (Chronic Obstructive Pulmonary Disease).
* History of unstable cardiovascular disease.
* BMI > 45
* Current use of anticoagulant medications.
* Upper Respiratory Infection (URI) within the previous 6 weeks
* Currently pregnant and/or unwillingness to practice medically acceptable birth control or complete abstinence during the study
* History of COVID-19 (coronavirus disease) in the past 6 months.

Protocol B:

Inclusion Criteria:

* Males or females between the ages 18 to 80 at the time of visit 1.
* Undergoing clinically indicated bronchoscopy for removal of mucus plugs.
* Clinical history of airway disease (including asthma, COPD and bronchiectasis) per patient report or medical record.
* Written informed consent obtained from subject.

Exclusion Criteria:

* Upper Respiratory Infection (URI) in the past 30 days.
* History of COVID-19 in the past 30 days.
* Currently pregnant during the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Change in FEV1 (Forced Expiratory Volume in the 1st second of Forced Expiration) | 1 week after and six months after research bronchoscopy.
  We will assess change from baseline FEV1 one week after and six months after removal of mucus plugs by bronchoscopy.
Incidence of Treatment-Emergent Adverse Events | Up to 1 week after the research bronchoscopy procedure.
  We will monitor the safety and tolerability of mucus plug removal by bronchoscopy by tracking the number of participants with treatment-related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: John Fahy, MD, MS, Principal Investigator — Professor of Medicine
Locations (1):
- UCSF Airway Clinical Research Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DUNNILL MS. The pathology of asthma, with special reference to changes in the bronchial mucosa. J Clin Pathol. 1960 Jan;13(1):27-33. doi: 10.1136/jcp.13.1.27. PMID 13818688